CLINICAL TRIAL: NCT06033014
Title: Clinical Implementation of a Novel Decision Support Tool in Patients With Ischemic Heart Disease
Acronym: PM Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Region Capital Denmark (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Henning Bundgaard, Professor of Cardiology, Consultant, MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: p-2023-14244
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The one-year mortality prediction, calculated by the PM Heart algorithm, will not be available to the physician.
- Intervention (Experimental): The one-year mortality prediction, calculated by the PM Heart algorithm, will be available to the physician.
  Interventions: Other: PM HeartIHD prediction

INTERVENTIONS:
Other: PM HeartIHD prediction — The calculated prediction and the explainability factors will be made available to the physician, which the physician then can decide to take into his/hers evaluation about further treatment.
  Arms: Intervention

SUMMARY:
The PM-Heart algorithm (PMHeartIHD) is an in-house developed software that predict the survival prognosis for the individual patient hospitalized with ischemic heart disease (IHD) after a coronary arteriography has been performed. The software is intended to be used as a clinical decision support system i.e. the calculated survival prognosis is expected to enhance the quality of the treating physician's therapeutic considerations concerning (minor) adjustments to the patients treatment and follow-up - all within the framework of the current medical guidelines. Thus, the algorithm does not "show the physician specifically what to do", but rather ensures a better knowledgebase for the overall interpretation and choice of management of the patient.

DETAILED DESCRIPTION:
To investigate the clinical usefulness of the developed clinical decision support system - the PMHeartIHD algorithm - we wish to investigate whether the clinical use of the algorithm will;

* Improve patient prognosis and,
* Minimize the risk of re-hospitalization,

compared to patients who are treated without the attending/treating physician knowing the algorithm's prognosis?

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients in one of the involved departments of cardiology (see below) with;
* Ischemic heart disease; the clinical presentation may be stable, worsening/unstable angina, non-ST-elevation myocardial infarction or ST-elevation myocardial infarction, and with - Significant coronary artery lesions or diffuse coronary artery disease on invasive coronary angiography during the admission

Exclusion Criteria:

* <18 years of age
* Living outside Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number and duration of readmissions within one month after randomization | From randomization to the study and up to 1 year hereafter
  A composite outcome of a) readmissions within one month, and 2) all-cause mortality within one year - for patients randomized to the study.
  All the outcomes listed below will be assessed as a comparison between the "intervention group" and the "control group".
Number and cause of death (all-cause mortality) within one year after randomization | From randomization to the study and up to 1 year hereafter
  A composite outcome of a) readmissions within one month, and 2) all-cause mortality within one year - for patients randomized to the study.

SECONDARY OUTCOMES:
Readmission(s) within 30 days of the randomization | Up to 30 days after randomization to the study.
  Readmission(s) within 30 days of the randomization. Incl. information on the quantity, duration, cause, outcome etc.
Cardiovascular readmission(s) within 30 days of the randomization | Up to 30 days after randomization to the study.
  Cardiovascular readmission(s) within 30 days of the randomization. Incl. information on the quantity, duration, cause, outcome etc.
Readmission(s) with acute coronary syndrome | From randomization to the study and up to 1 year hereafter
  Readmission(s) with acute coronary syndrome. Incl. information on the quantity, duration, cause, outcome etc.
One-year survival | From randomization to the study and up to 1 year hereafter
  One-year survival
Total number of days the primary hospitalization lasts | From randomization to the study and up to 1 year hereafter
  Length (i.e. total number of days) of the primary hospitalization (i.e. when the patient is randomized to the study).
Total number of days at the hospital incl. hospitalizations during the first year after inclusion | From randomization to the study and up to 1 year hereafter
  Total number of days in hospital during the first year after inclusion
Number of hospitalizations the first year | From randomization to the study and up to 1 year hereafter
  Number of hospitalizations the first year
Number and type of performed cardiac investigations | From randomization to the study and up to 1 year hereafter
  Number and type of performed cardiac investigations; i.e. TTE, KAG, Heart-CT, Holter/R-tests, ECG, blood samples, etc.
Number of cardiac follow-up consultations at the hospital | From randomization to the study and up to 1 year hereafter
  Number of cardiac follow-up consultations at the hospital
Number of check-ups for cardiovascular reasons at the general practitioner | From randomization to the study and up to 1 year hereafter
  Number of check-ups for cardiovascular reasons at the general practitioner.
Number of cardiovascular drugs at discharge | From randomization to the study and up to 1 year hereafter
  Number of cardiovascular drugs at discharge + after 1 year.
Dosages (DDD) of drugs at discharge | Up to 1 year after randomization to study.
  Dosages (DDD) of drugs at discharge + after 1 year.
Incidence of a) new ischemic events, b) arrhythmias, c) and/or heart failure | Up to 1 year after randomization to study.
  Incidence of a) new ischemic events, b) arrhythmias, c) and/or heart failure
Health economic analyses of implementing the algorithm | Up to 1 year after randomization to study.
  Health economic analyses: How does implementing the algorithm alter the overall costs and resource spending, incl. e.g. social benefits, compared with standard-of-care.
  i.e. does knowing a more precise 1-year mortality prediction reduce/increase the resource consumption.
  Will be based on economic analyses of the costs related to the abovementioned outcome measurements.
The algorithm's reception and introduction in clinical use | Before start of clinical study and up to 1 year after randomization to study.
  We wish to investigate how the algorithm is introduced and received in the clinic, both by the medical staff but also the patients.
  Will be investigated using interviews.
The usability of the algorithm | Before start of clinical study and up to 1 year after randomization to study.
  The usability of the algorithm i.e. is it easy to use/understand, any praise or criticisms, ideas for new features etc.
  Will be based on questionaires and feedback from users.
How, and to what extend, is the algorithm used by the medical staff. | Before start of clinical study and up to 1 year after randomization to study.
  We wish to investigate how, and to what extend, the algorithm is used by the medical staff, e.g. are the medical staff inclined to use the prediction, does it alter their treatment choices etc.
  Will be based on questionaires, interviews, feedback from users, and assessment of "look-ups".

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, The Heart Centre, Rigshospitalet Copenhagen University Hospital., Copenhagen Ø, Denmark